CLINICAL TRIAL: NCT06666868
Title: CARD (Comfort Ask Relax Distract) for Community-based Pharmacy Vaccinations - Phase 2
Brief Title: CARD for Community Pharmacy Vaccinations - Phase 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Wholehealth Pharmacy Partners (Unknown)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43097-2024
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Vaccination; Vaccination Pain; Vaccination Reaction; Vaccination Pharmacy
Keywords: vaccination reaction; vaccination experience

STUDY DESIGN:
Intervention Model Description: Cluster trial involving at least 8 community pharmacies allocated in a 1:1 ratio to: 1) repeat use or 2) first-time use of the CARD system for vaccination delivery in 2024-2025 fall/winter vaccination season.
Who Masked: Participant, Outcomes Assessor
Masking Description: Vaccine clients are blinded to the hypothesis. Providers are aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sustained CARD (Experimental): CARD is being used for the 2nd year in a row as the vaccination delivery framework in participating pharmacies (It was used in the 2023-2024 fall/winter vaccination season and is now being sustained in the 2024-2025 fall/winter season). CARD comprises of education, environment, engagement and evaluation components.
  Interventions: Behavioral: Sustained CARD
- First-time CARD (Active Comparator): CARD is being used for the 1st time as the vaccination delivery framework in participating pharmacies (2024-2025 fall/winter vaccinations only). CARD comprises of education, environment, engagement and evaluation components.
  Interventions: Behavioral: First-time CARD

INTERVENTIONS:
Behavioral: Sustained CARD — This group is using CARD for the 2nd year in a row in participating pharmacies as the vaccination delivery framework (It was used in the 2023-2024 fall/winter vaccination season and is now being sustained in the 2024-2025 fall/winter vaccination season).
  Other Names: Sustained CARD use
  Arms: Sustained CARD
Behavioral: First-time CARD — CARD is being used for the 1st time in participating pharmacies as the vaccination delivery framework (2024-2025 fall/winter vaccination season).
  Other Names: First-time CARD use
  Arms: First-time CARD

SUMMARY:
This study is phase 2 of a cluster trial integrating the CARD (Comfort Ask Relax System) in community pharmacies affiliated with Wholehealth Pharmacy Partners. It involves continuing CARD in pharmacies randomized to CARD in phase 1 of the trial (2023-2024 fall/winter vaccination season), and initiating CARD in pharmacies randomized to Control (usual care) in phase 1 of the trial. Both groups will use CARD for delivery of vaccinations during the 2024-2025 fall/winter vaccination season.

DETAILED DESCRIPTION:
This study is a continuation of a previous cluster trial. Pharmacies that participated in the original trial will be asked if they want to volunteer for the present study. They will all use the CARD system as the vaccination delivery system for their community pharmacies during the 2024-2025 fall/winter vaccination season. They will collect feedback from vaccine clients using a paper survey that tracks experiences, including symptoms, during vaccination. The responses will be compared between groups.

The sample size is limited by the number of pharmacies that volunteer. We expect 8 pharmacies will participate in a 1:1 ratio (about 1/3 of all pharmacies in original cluster trial), with a total of at least 500 vaccination clients. We will collect data for all vaccinations that are conducted and for which client feedback data are available. Thus, the sample size is expected to deviate from the estimated sample size of 500.

ELIGIBILITY:
Inclusion Criteria:

* clients undergoing vaccination in participating pharmacies and providers working in participating pharmacies

Exclusion Criteria:

* able to speak and write in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Experience with vaccination | Within 15 minutes of vaccination
  Self-reported experience about how much CARD helped (4-point Likert scale and dichotomized)

SECONDARY OUTCOMES:
Pain | Within 15 minutes of vaccination
  Self-reported pain during vaccination (0-10)
Fear | Within 15 minutes of vaccination
  Self-reported fear during vaccination (0-10)
Dizziness | Within 15 minutes of vaccination
  Self-reported dizziness during vaccination (0-10)
Fainting | Within 15 minutes of vaccination
  Self-reported fainting during vaccination (yes/no) confirmed by provider
Overall experience | Within 15 minutes of vaccination
  Self-reported overall experience (5-point Likert scale, and dichotomized)
Vaccination decision-making | Within 15 minutes of vaccination
  Self-reported vaccination decision-making (5-point Likert scale, and dichotomized)
Implementation outcomes | Within 3 months of vaccination season ending
  Provider quantitative and qualitative feedback on surveys and interviews (assessing implementation outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — Leslie Dan Faculty Of Pharmacy, University Of Toronto
Locations (1):
- Leslie Dan Faculty of Pharmacy, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not have permission to share individual participant data.